CLINICAL TRIAL: NCT02516969
Title: A Prospective, Randomized Phase II Study of Surgery With or Without Adjuvant Stereotactic Body Radiotherapy (SBRT) in Patients With Previously-Irradiated Head and Neck Cancer
Brief Title: Surgery With or Without Adjuvant Stereotactic Body Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A. Clump, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David A. Clump, MD, PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-151
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Cancer
Keywords: Stereotactic Body Radiotherapy (SBRT)
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic Body Radiotherapy (Experimental): Subjects will receive Stereotactic Body Radiotherapy at the following levels: Treatment Volumes <25cc will receive 40Gy (5 fractions of 8Gy per fraction) or treatment Volumes ≥25cc will receive 44-50Gy (5 fractions of 8.8-10Gy per fraction). Ideally all tumors volumes ≥25cc will receive 50Gy over 5 fractions, however at the discretion of the treating radiation oncologist based on tumor bed volume, prior radiation dose, and proximity to critical organs the dose can be reduced to 44Gy over 5 fractions as outlined in prior SBRT protocols.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Radiation
  Other Names: SBRT

SUMMARY:
Comparison of patients with operable, recurrent previously-irradiated squamous cell head-and-neck cancers with or without adjuvant SBRT.

DETAILED DESCRIPTION:
This study aims to determine prognostic factors that may predict the likelihood of local failure, regional failure, to guide future management, to compare the impact of adjuvant SBRT versus a wait-and-see approach on patient reported quality of life (PR-QoL), and to compare surgical versus SBRT-induced immunological serum markers in relation to local control. Recruitment includes patients with recurrent or second-primary head-and-neck squamous cell carcinomas within a previously-irradiated field with high-risk features compromised/positive surgical margins or extra-nodal extension) following macroscopic complete (R0/R1) salvage surgery.

Participants receive Stereotactic Body Radiotherapy at the following levels:

Treatment Volumes <25cc will receive 40Gy (5 fractions of 8Gy per fraction) or treatment Volumes ≥25cc will receive 44-50Gy (5 fractions of 8.8-10Gy per fraction). Ideally all tumors volumes ≥25cc will receive 50Gy over 5 fractions, however at the discretion of the treating radiation oncologist based on tumor bed volume, prior radiation dose, and proximity to critical organs the dose can be reduced to 44Gy over 5 fractions as outlined in prior SBRT protocols. Evaluations to compare the efficacy of adjuvant SBRT versus wait-and-see, include Local Control, Regional and distant control, Progression-free survival, Overall survival and Patient-Reported Quality-of-Life (PR-QoL).

Evaluations conducted to assess the safety of adjuvant SBRT following salvage surgery include recording of all toxicity data per National Cancer Institute Common Toxicity Criteria Events Scale version 4.0 and prospectively administering the previously-validated University of Washington Quality-of-Life-Revised (UW-QoL-R) questionnaire measuring patient-reported quality-of-life (PR-QoL).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven recurrent or second-primary head-and-neck cancer receiving prior radiotherapy with or without chemotherapy.
* Prior radiotherapy to a dose of ≥50Gy
* No evidence of distant metastases
* Macroscopic complete salvage surgery with curative intent (surgery was not performed only for biopsy or palliation). Final pathology and imaging must indicate a R0 or R1 resection (no gross disease remaining).
* High-risk pathologic features must be present: compromised/positive surgical margins (≤ 2mm) or extra-nodal extension (patient with other high-risk features gross perinueral invasion, bone invasion, angiolyphatic invasion, or a constellation of these factors may be eligible based on case-by-case basis at discretion of principal investigator).
* Karnofsky Performance Status ≥60 (ECOG 0-2)
* Any number or type of prior chemotherapy is allowed (patient may receive concurrent or adjuvant systemic therapy such as cetuximab at the discretion of the treating oncologic team)

Exclusion Criteria:

* Evidence of distant metastases on any staging or imaging modality
* Women who are breast feeding, or have a positive pregnancy test (reproductive age should use effective birth control during study if randomized to SBRT treatment arm)
* Any patient with gross residual disease following salvage surgery
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08; Primary Completion 2019-05-30 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiotherapy: Stereotactic Body Radiotherapy at the following levels: Treatment Volumes <25cc will receive 40Gy (5 fractions of 8Gy per fraction) or treatment Volumes ≥25cc will receive 44-50Gy (5 fractions of 8.8-10Gy per fraction). Ideally all tumors volumes ≥25cc will receive 50Gy over 5 fractions, however at the discretion of the treating radiation oncologist based on tumor bed volume, prior radiation dose, and proximity to critical organs the dose can be reduced to 44Gy over 5 fractions as outlined in prior SBRT protocols.
- Observation: No Stereotactic Body Radiotherapy
Period: Overall Study
Arm/Group | Stereotactic Body Radiotherapy | Observation
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients participating in the trial.
Groups:
- Observation Cohort: No Stereotactic Body Radiotherapy
- Total: Total of all reporting groups
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [58.00 to 67.00] | 64 [58.00 to 71.50] | 63 [58 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Karnofsky Performance Status (KPS) [Median (Inter-Quartile Range); unit: score on a scale] — The Karnofsky Performance Status (KPS) scores range 0 - 100. Higher KPS scores means the patient is better able to carry out daily activities, used to determine a patient's prognosis, and used to measure changes in a patient's overall ability to function.
  score on a scale | 80.0 [60.00 to 80.00] | 80.0 [80.00 to 85.00] | 80.0 [80.0 to 80.0]

OUTCOME MEASURES:

1. Primary Outcome: 1-year Local Control
Description: Local progression-free-survival (LPFS) is the number of months from the initiation of study treatment until (local) progression of disease or death from any cause. Progression is defined as the appearance of a new metastatic lesion or objective tumor progression. Clinically detected lesions will only be considered measurable when superficial (vis-à-vis skin modules and palpable lymph nodes). The lesion must be accurately measured in at least one dimension ≥ 10mm. Methods for measuring disease status include CT, PET/CT or MRI.
Time Frame: Up to 1 year
Population: Patients with/without SBRT treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Observation Cohort: No Stereotactic Body Radiotherapy treatment
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Median survival is not reached. Insufficient number of participants with event of (local) progression. | NA [2 to NA] — Upper bound of 95% CI not available. Insufficient number of participants with event of (local) progression.

2. Secondary Outcome: Number of Participants With Acute Toxicities of Adjuvant SBRT
Description: Toxicities are assess according to the National Cancer Institute Common Toxicity Criteria Events Scale (CTCAE), v4. Acute toxicities are those seen within 3 months of completion of Stereotactic Body Radiotherapy. Toxicity in patients is documented immediately prior to randomization and 8-12 weeks post-treatment. Adverse events are Grade 1 and 2 and Serious Adverse events are Grade 3 and 4 events.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
Participants
  Grade 3 - Oral Mucositis | 1 | 0
  Grade 1 Dysphagia | 1 | 1
  Grade 1 Dysphonia | 1 | 0
  Grade 1 Edema | 1 | 0
  Grade 1 Fatigue | 1 | 1
  Grade 1 Lymphedema | 1 | 1
  Grade 1 Odynophagia | 1 | 0
  Grade 1 Pain | 1 | 0
  Grade 1 Radiation Dermatitis | 1 | 0
  Grade 1 Xerostomia | 1 | 1
  Grade 2 Xerostomia | 1 | 0
  Grade 2 Pain | 1 | 0
  Grade 1 Dysgeusia | 0 | 1
  Grade 2 Fibrosis | 0 | 1
  Grade 1 Jaw Pain | 0 | 1
  Grade 1 Otalgia | 0 | 1
  Grade 1 telangiectasia | 0 | 1
  Grade 1 Trismus | 0 | 1

3. Secondary Outcome: Number of Participants With Late Toxicities of Adjuvant SBRT
Description: Toxicities will be assessed according to the National Cancer Institute Common Toxicity Criteria Events Scale (CTCAE), v4. Late toxicities will be those seen after 3 months of completion of Stereotactic Body Radiotherapy. Adverse events are Grade 1 and 2 and Serious Adverse events are Grade 3 and 4 events.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
Participants
  Grade 3 Pneumonia | 1 | 0
  Grade 1 Aspiration | 2 | 0
  Grade 1 Dysgeusia | 2 | 0
  Dysphagia | 1 | 0
  Grade 1 Fatigue | 1 | 0
  Grade 1 Fibrosis | 1 | 0
  Grade 2 Fibrosis | 1 | 0
  Grade 2 Infection (Thrush) | 1 | 0
  Grade 1 Lymphedema | 1 | 0
  Grade 2 Lymphedema | 1 | 0
  Grade 2 Pain | 1 | 0
  Grade 1 Trismus | 1 | 0
  Grade 2 Ulceration | 1 | 0
  Grade 1 Xerostomia | 1 | 0
  Grade 2 Xerostomia | 1 | 0

4. Secondary Outcome: Progression-free Survival (PFS) Locoregional
Description: LRPFS is defined as the time from the date of randomization to the date of local or regional recurrence, whichever occurs first, or the date of death from any cause. Subjects who are alive and have not progressed will be censored at their last follow-up date. Progression is defined as the appearance of a new metastatic lesion or objective tumor progression. Clinically detected lesions will only be considered measurable when superficial (vis-à-vis skin modules and palpable lymph nodes). The lesion must be accurately measured in at least one dimension ≥ 10mm. Methods for measuring disease status include CT, PET/CT or MRI.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Median LRPFS not reached. The 95% CI not available. Insufficient number of participants with event of (locoregional) progression. | NA [2 to NA] — Median LRPFS not reached. Upper bound of 95% CI not available. Insufficient number of participants with event of (locoregional) progression.

5. Secondary Outcome: Progression-free Survival (DPFS) Distant
Description: Distant progression-free-survival (DPFS) is the time from the date of randomization to the date of distant progression or the date of death from any cause. Progression is defined as the appearance of a new metastatic lesion or objective tumor progression. Clinically detected lesions will only be considered measurable when superficial (vis-à-vis skin modules and palpable lymph nodes). The lesion must be accurately measured in at least one dimension ≥ 10mm. Methods for measuring disease status include CT, PET/CT or MRI.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Median DPFS not reached. The 95% CI not available. Insufficient number of participants with event of (distant) progression. | NA [11 to NA] — Median DPFS not reached. Upper bound of 95% CI not available. Insufficient number of participants with event of (distant) progression.

6. Secondary Outcome: Overall Progression Free Survival (PFS)
Description: Overall progression free survival is the total of the three survival time measurements; PFS = local + regional + distant. Progression is defined as the appearance of a new metastatic lesion or objective tumor progression. Clinically detected lesions will only be considered measurable when superficial (vis-à-vis skin modules and palpable lymph nodes). The lesion must be accurately measured in at least one dimension ≥ 10mm. Methods for measuring disease status include CT, PET/CT or MRI.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Median survival not reached. The 95% CI not available. Insufficient number of participants with event of progression. | NA [2 to NA] — Median survival not reached. Upper bound of 95% CI not available. Insufficient number of participants with event of progression.

7. Secondary Outcome: Overall Survival (OS)
Description: The overall survival time is the measurement of time between the date of randomization and death from any cause.
Time Frame: Up to 5 years
Population: Patients with/without SBRT treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Observation: No Stereotactic Body Radiotherapy treatment
Arm/Group | Stereotactic Body Radiotherapy | Observation
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Median OS not reached. 95% CI was not available. Insufficient number of participants with event of death. | NA [NA to NA] — Median OS not reached. 95% CI was not available. Insufficient number of participants with event of death.

8. Secondary Outcome: Quality of Life (UW-QoL-R)
Description: The University of Washington Quality of Life questionnaire (revised) is a self-administered 16 item inquiry given to patients with head and neck cancer. The first 12 items ask the patient to score domains (such as pain, appearance, swallowing) from 0 (worse) to 100 (best). The arithmetic mean is then computed, yielding one number between 0 and 100. The higher the number, the "better" the patient is considered to be faring. The item simply asks the patient to choose the top 3 issues which have been bothering the patient over the past 7 days. The issues include physical symptoms, emotions and appearance. The final 3 questions provide a global assessment by asking the patient to consider their overall well-being over the past 7 days and provide possible answers ranging from excellent to very poor. For trial analysis: Period=1: before surgery, Period=2: after surgery, but before SBRT for patients in the SBRT arm, Period=3: after SBRT.
Time Frame: Up to 2 years
Population: Patients with/without SBRT treatment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Stereotactic Body Radiotherapy | Observation
Number analyzed (Participants) | 3 | 4
score on a scale
  Period 1: Pain | 100.00 [100.00 to 100.00] | 75.00 [75.00 to 75.00]
  Period 2: Pain | 100.00 [100.00 to 100.00] | 75.00 [37.50 to 100.00]
  Period 3: Pain | 75.00 [50.00 to 75.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Appearance | 75.00 [75.00 to 75.00] | 75.00 [75.00 to 75.00]
  Period 2: Appearance | 50.00 [50.00 to 50.00] | 87.50 [50.00 to 100.00]
  Period 3: Appearance | 75.00 [62.50 to 100.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Activity | 50.00 [50.00 to 50.00] | 75.00 [75.00 to 75.00]
  Period 2: Activity | 50.00 [50.00 to 50.00] | 75.00 [62.50 to 87.50]
  Period 3: Activity | 62.50 [62.50 to 75.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Recreation | 62.50 [50.00 to 75.00] | 75.00 [75.00 to 75.00]
  Period 2: Recreation | 25.00 [25.00 to 25.00] | 75.00 [62.50 to 87.50]
  Period 3: Recreation | 62.50 [62.50 to 75.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Swallowing | 67.00 [67.00 to 67.00] | 67.00 [67.00 to 67.00]
  Period 2: Swallowing | 67.00 [67.00 to 67.00] | 67.00 [33.50 to 83.50]
  Period 3: Swallowing | 67.00 [67.00 to 67.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Chewing | 50.00 [0.00 to 100.00] | 100.00 [100.00 to 100.00]
  Period 2: Chewing | 50.00 [50.00 to 50.00] | 75.00 [50.00 to 100.00]
  Period 3: Chewing | 50.00 [50.00 to 100.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Speech | 75.25 [67.00 to 83.50] | 67.00 [67.00 to 67.00]
  Period 2: Speech | 33.00 [33.00 to 33.00] | 100.00 [100.00 to 100.00]
  Period 3: Speech | 67.00 [66.50 to 100.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Shoulder | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Period 2: Shoulder | 100.00 [100.00 to 100.00] | 100.00 [83.50 to 100.00]
  Period 3: Shoulder | 67.00 [66.50 to 100.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Taste | 50.00 [33.00 to 67.00] | 67.00 [67.00 to 67.00]
  Period 2: Taste | 33.00 [33.00 to 33.00] | 67.00 [50.00 to 83.50]
  Period 3: Taste | 67.00 [50.00 to 67.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Saliva | 50.00 [33.00 to 67.00] | 67.00 [67.00 to 67.00]
  Period 2: Saliva | 0.00 [0.00 to 0.00] | 83.50 [50.00 to 100.00]
  Period 3: Saliva | 67.00 [33.00 to 76.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Mood | 75.00 [75.00 to 75.00] | 75.00 [75.00 to 75.00]
  Period 2: Mood | 50.00 [50.00 to 50.00] | 75.00 [50.00 to 75.00]
  Period 3: Mood | 75.00 [75.00 to 75.00] | NA [NA to NA] — Survey not completed by patient(s).
  Period 1: Anxiety | 83.50 [67.00 to 100.00] | 67.00 [67.00 to 67.00]
  Period 2: Anxiety | 67.00 [67.00 to 67.00] | 67.00 [50.00 to 83.50]
  Period 3: Anxiety | 100.00 [67.00 to 100.00] | NA [NA to NA] — Survey not completed by patient(s).

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Adverse events are Grade 1 and 2 and Serious Adverse events are Grade 3 and 4 events per National Cancer Institute Common Toxicity Criteria Events Scale (CTCAE), v4.
Arm/Group | Stereotactic Body Radiotherapy | Observation Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiotherapy (N=3) | Observation Cohort (N=4)
Oral Mucositis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiotherapy (N=3) | Observation Cohort (N=4)
Dysphagia (Gastrointestinal disorders) | 2 | 1
Dysphonia (Investigations) | 1 | 0
Edema (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Lymphedema (Vascular disorders) | 3 | 1
Odynophagia (Investigations) | 1 | 0
Pain (General disorders) | 3 | 1
Radiation Dermatitis (Injury, poisoning and procedural complications) | 1 | 0
Xerostomia (Gastrointestinal disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Fibrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Otalgia (Ear and labyrinth disorders) | 0 | 1
telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Infection (Thrush) (Infections and infestations) | 1 | 0
Ulceration (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02516969/Prot_SAP_000.pdf